CLINICAL TRIAL: NCT02674438
Title: Comparison of Outcomes and Access to Care for Heart Failure Trial
Acronym: COACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Douglas Lee, Senior Scientist, Institute for Clinical Evaluative Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Intervention (Experimental): Two components to the intervention: (1) clinical algorithm for prognostication, and (2) post-discharge follow-up in the RAPID-HF clinic
  Intervention #1 - Clinical algorithm: the EHMRG30-ST risk score which will be used to categorize patients as high, intermediate, or low risk. The clinical algorithm will be used to guide clinicians to decide on admission to hospital, observation during a short stay hospital admission (3 days or less), or emergency department discharge.
  Intervention #2 - Referral to RAPID-HF (Rapid Ambulatory Program for Investigation and Diagnosis of HF) transitional care clinic: visit to RAPID-HF within 48-72 hours of discharge. Care provided in RAPID-HF by cardiologist + nurse for up to 30 days from date of discharge.
  Interventions: Other: Risk stratification and transitional care intervention
- Control (No Intervention): Usual care without access to the EHMRG30-ST scoring system, decision algorithm, or RAPID-HF clinic.

INTERVENTIONS:
Other: Risk stratification and transitional care intervention — Intervention consists of 2 components:
  1. Risk stratification: Determination of risk using the EHMRG 7-day and 30-day risk scores (EHMRG30-ST), where decision to admit, observe, or discharge the patient will be guided by the result of the risk scores
  2. Transitional care: Follow-up care in the RAPID-HF transitional care clinic begins at 48-72 hours after emergency department or hospital discharge. Care provided by cardiologist + nurse for up to 30 days after emergency department or hospital discharge.
  Arms: Active Intervention

SUMMARY:
Heart failure is a condition where the heart pump does not function normally causing the lungs to become congested. The primary symptom of heart failure is shortness of breath, and this often leads to patients visiting the emergency department for care. Decision-making in the emergency department is a high-stakes situation, where there is a need for decision support to guide clinicians to make better decisions about admission to hospital or discharge home. Many low-risk patients who could potentially be managed at home are admitted to hospital whereas some patients who are thought safe to discharge are actually high risk and will have adverse outcomes if they are discharged home from the emergency department.

In this trial, the investigators will study a new strategy for heart failure care, comprised of a computer algorithm to help doctors make decisions in the emergency department about the risk of their patient. For low-risk patients who are discharged home from the emergency department or after a short hospital stay, patients will be referred to a rapid follow-up clinic where the heart specialist team will rapidly assess and treat patients.

DETAILED DESCRIPTION:
Overview: Randomized intervention trial to examine the impact of an acute heart failure strategy, which incorporates risk stratification and rapid outpatient care after discharge.

Study Population: Patients presenting to the emergency department with heart failure will be eligible for study inclusion.

Inclusion and Exclusion Criteria for the Study:

1. Age 18 years or older
2. Presents to the emergency department with acute heart failure diagnosed clinically and verified by a primary diagnosis of heart failure (ICD-10-CA code I50) on the emergency department facesheet.

Exclusion criteria:

1. Does not meet Framingham criteria for heart failure
2. Heart failure diagnosis unlikely according to B-type natriuretic peptide values

   1. BNP <100 pg/mL or
   2. NT-proBNP <300 pg/mL
3. End stage renal disease on dialysis
4. Palliative patient with do not resuscitate (DNR) order present prior to emergency department arrival
5. Limited mobility to attend outpatient clinic visits
6. Dementia
7. Nursing home resident
8. No permanent home address
9. Non-resident of Ontario
10. Self-discharge from emergency department
11. Invalid Ontario health insurance number

Inclusion and Exclusion Criteria for the RAPID-HF Clinic:

Inclusion criteria:

1. Patients with heart failure presenting to the emergency department meeting overall study eligibility criteria
2. Discharged at any time within the first 3 days after emergency department presentation
3. Using the EHMRG30-ST risk score:

   1. Any low-risk patient who is able to be discharged within 3 days of initial emergency department presentation
   2. Some intermediate-to-low risk zone EHMRG30-ST may be eligible if judged to be clinically stable
4. Patient agrees to be discharged early from either the emergency department or hospital
5. Able to attend outpatient clinic visits

Exclusion criteria:

1. High risk zone of EHMRG30-ST
2. Pre-cardiac transplant
3. Active cardiac ischemia without diagnostic testing done during hospital stay
4. Uncontrolled arrhythmia
5. Worsening renal failure compared to baseline renal function
6. Significant abnormality of vital signs at the time of referral:

   1. Oxygen saturation on room air less than or equal to 90% which is not usual for patient
   2. Systolic blood pressure < 90 mmHg with symptoms of hypotension
   3. Heart rate in sinus rhythm greater than or equal to 100 bpm
   4. Respiratory rate > 20 breaths/minute
7. New heart failure diagnosis (not an absolute contraindication to referral, but not recommended)

Intervention: The study involves 2 components: clinical algorithm for prognostication and post-discharge follow-up in the Rapid Ambulatory Program for Investigation and Diagnosis of Heart Failure (RAPID-HF) clinic.

The clinical decision-support algorithm intervention is a composite of 7-day and 30-day risk calculator (called EHMRG30-ST). Using the EHMRG30-ST algorithm, patients will be categorized as high, intermediate, or low risk. The decision support algorithm will recommend hospital admission or discharge/observation based on patient risk to assist clinicians making the final decision to admit or discharge. Low risk patients may be discharged early (within 3 days of initial presentation) and referred to the RAPID-HF clinic.

Patients referred to RAPID-HF will be assessed ideally within 48-72 hours of discharge. RAPID-HF provides transitional care for up to 30 days after discharge. After 30-days, care is transferred to primary care provider or specialist for ongoing care.

Study Design: Using a stepped-wedge design, participating sites will be randomized to the active intervention. At each step, hospitals that have not yet been randomized will serve as control sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to an emergency department with heart failure

Exclusion Criteria:

* Palliative or DNR
* Dialysis dependent
* Non-Ontario resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5452 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Co-primary outcome: 30 day early events | 30 days
  Time to composite of death or cardiovascular hospitalization (nonelective, los > 1 day)
Co-primary outcome: 20 month extended events | 20 month follow-up
  Time to composite of death or cardiovascular hospitalization (nonelective, los > 1 day)

SECONDARY OUTCOMES:
All-cause death | 30 days
  Time to death
Cardiovascular hospitalization | 30 days
  Time to cardiovascular hospitalization (nonelective, los > 1 day)
Heart failure hospitalization | 30 days
  Time to heart failure hospitalization (nonelective, los > 1 day)
All-cause death | 20 months
  Time to death (nonpalliative)
Cardiovascular hospitalization | 20 months
  Time to cardiovascular hospitalization (nonelective, los > 1 day)
Heart failure hospitalization | 20 months
  Time to heart failure hospitalization (nonelective, los > 1 day)

OTHER OUTCOMES:
Patient-centered outcome | 1) 30-day and 2) 20 month
  Time to nonelective emergency department visit (CTAS 1-4), death or cardiovascular hospitalization
Early discharge | 3 days
  Proportion of patients discharged within 3 days of emergency presentation

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lee, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Genera Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Due to Ontario privacy regulations, unable to share data

REFERENCES:
- [Derived] Lee DS, Straus SE, Farkouh ME, Austin PC, Taljaard M, Chong A, Fahim C, Poon S, Cram P, Smith S, McKelvie RS, Porepa L, Hartleib M, Mitoff P, Iwanochko RM, MacDougall A, Shadowitz S, Abrams H, Elbarasi E, Fang J, Udell JA, Schull MJ, Mak S, Ross HJ; COACH Trial Investigators. Trial of an Intervention to Improve Acute Heart Failure Outcomes. N Engl J Med. 2023 Jan 5;388(1):22-32. doi: 10.1056/NEJMoa2211680. Epub 2022 Nov 5. PMID 36342109